CLINICAL TRIAL: NCT06288516
Title: BenRalizumab Effect on Airway Remodeling in Severe Eosinophilic asTHmatics
Brief Title: BenRalizumab Effect on Airway Remodeling in Severe asTHma
Acronym: BREATH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Pulmonary Clinic, University of Ioannina (Unknown); Pulmonary Clinic, Democritus University of Thrace (Unknown); 2nd Pulmonary Clinic, Kapodistrian University of Athens (Unknown); University Hospital of Crete (Other); Pulmonary and Respiratory Failure Department, National and Kapodistrian University of Athens (Unknown); University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Kalliopi Domvri, Academic Fellow in the laboratory of Histology-Embryology, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7484
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Asthma; Eosinophilic; Airway Remodeling
Keywords: severe asthma; airway remodeling; eosinophilic; biomarkers; bronchoscopy
MeSH Terms: conditions — Pulmonary Eosinophilia; Airway Remodeling; Asthma | interventions — benralizumab; Biological Products

STUDY DESIGN:
Intervention Model Description: Benralizumab (30mg) administered subcutaneously every 4 weeks for the first 3 dose and then every 8 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benralizumab Arm A (Experimental): Benralizumab (30mg) administered subcutaneously every 4 weeks for the first 3 dose and then every 8 weeks.
  Interventions: Drug: Benralizumab 30 mg/ml
- No intervention Arm B (No Intervention): No intervention. Standard of care as treatment.

INTERVENTIONS:
Drug: Benralizumab 30 mg/ml — Benralizumab administered subcutaneously every 4 weeks for the first 3 dose and then every 8 weeks
  Other Names: biological
  Arms: Benralizumab Arm A

SUMMARY:
Response to biologic therapies in severe asthma is variable, with patients being either non-responders, responders or super-responders. There is currently no explanation for this broad variation in response. It is important to examine whether these patients have distinct characteristics that could help the treating physician in making the correct diagnosis in clinical practice.

Aim of this clinical study is to evaluate the efficacy of benralizumab, a humanized an anti-interleukin 5 receptor α monoclonal antibody in patients with severe eosinophilic asthma and to evaluate airway remodeling before and after benralizumab treatment.

Hypothesis Identification of pathological and clinical characteristics in patients with severe eosinophilic asthma after benralizumab treatment regarding the airway remodeling, inflammatory cells, and other biomarkers on a long-term basis.

Research questions Is there any improvement in airway remodeling? Are there any biomarkers to predict response to benralizumab treatment in severe eosinophilic asthmatic patients?

DETAILED DESCRIPTION:
Interleukin (IL)-5 is the main cytokine responsible for the activation of eosinophils, hence therapeutic strategies have been investigated and developed for clinical use. Biologics targeting IL-5 and its receptor have been recently approved and used as add-on therapy for severe eosinophilic asthma resulting in a reduction in the circulating eosinophil count, improvement in lung function and exacerbation reduction in patients with severe asthma.

Response to biologic therapies in severe asthma is variable, with patients being either non-responders, responders or super-responders. There is currently no explanation for this broad variation in response. It is important to examine whether these patients have distinct characteristics that could help the treating physician in making the correct diagnosis in clinical practice.

Aim of this clinical study is to evaluate the efficacy of benralizumab, a humanized an anti-interleukin 5 receptor α monoclonal antibody in patients with severe eosinophilic asthma and to evaluate airway remodeling before and after benralizumab treatment. Every patient will be a control to himself by comparing baseline's biomarker measurements of each patient to the following timepoint's measurements. However, we have added 10 severe asthmatics with no intervention, receiving standard of care as control groups to make more comparisons.

Several methods are used to investigate airway inflammation: direct measurements (like bronchial biopsies or bronchoalveolar lavages) and indirect methods (like symptom assessment, blood sample analysis and lung function tests). The direct techniques have the advantage of reliably assessing the airway inflammation, but they are invasive and not feasible at large scale because of patient discomfort and the risk incurred. As for the indirect methods, they poorly correlate with the direct assessment of airway inflammation.

In this study, among patients' clinical characteristics spirometry, biomarkers of inflammation such as blood eosinophils, Fractional Exhaled Nitric Oxide (FeNO), immunoglobulin E (IgE) levels), and airway remodeling via bronchoscopy will be evaluated. The precise effects of increased airway smooth muscle area on airway narrowing are not known and may vary with disease severity. In addition, biomarkers of inflammation will also be evaluated before and after 52-week of benralizumab treatment in biological fluids (serum and bronchial samples). Biomarkers of inflammation are very important to identify treatment response.

Besides, asthmatic disease is characterized by a chronic mucosal inflammatory process, which results in irreversible changes of the bronchial wall, known today as "bronchial remodeling". Glandular and smooth muscle fibers hyperplasia and/or hypertrophy, goblet cells hyperplasia, and variable thickening of basement membrane (BM) present under the respiratory epithelium are part of these morphological changes. the changes generated at the epithelium-connective interface account for an "adaptive response" to inflammatory stress and sporadic bronchoconstriction. However, current data on BM reactivity in asthmatic patient are still incomplete for an accurate assessment of its involvement in pathogenesis and specifically in bronchial wall remodeling, mainly as collagen deposits in lamina reticularis are not correlated to the degree of disease severity.

Moreover, it is increasingly evident that severe asthma is not a single disease, as evidenced by the variety of clinical presentations, physiologic characteristics, and outcomes seen in patients with asthma. To better understand this heterogeneity, the concept of asthma phenotyping and endotyping has emerged. Phenotyping integrates both biological and clinical features, from molecular, cellular, morphologic, and functional to patient-oriented characteristics with the goal to improve therapy. Ultimately, these phenotypes evolve into asthma "endotypes," which combine clinical characteristics with identifiable mechanistic pathways. Biomarkers, defined as characteristics that can be objectively measured and serve as an indicator of underlying biological processes or pathogenesis, are crucial in defining phenotypes and endotypes. In asthma, genetic polymorphisms, measures of airway physiology, and levels of inflammatory mediators in urine, blood, sputum, tissue, exhaled gas, and breath condensate have all been studied as potential markers to improve and objectify asthma diagnosis and management. Developing such tools will allow us to phenotype and endotype the various clinical patterns described in asthma, with the ultimate goal of tailoring therapy based on a specific biomarker profile. Biomarkers can then be used to help better understand the pharmacologic response to an intervention and adjust therapy accordingly.

Biomarkers have been critical for studies of disease pathogenesis and the development of new therapies in severe asthma. In particular, biomarkers of type 2 inflammation have proven valuable for endotyping and targeting new biological agents. Because of these successes in understanding and marking type 2 inflammation, lack of knowledge regarding non-type 2 inflammatory mechanisms in asthma will soon be the major obstacle to the development of new treatments and management strategies in severe asthma. Other potential biomarkers include innate lymphoid cells, IL-33 or thymic stromal lymphopoietin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained at screening visit, before any assessment will be performed. Subjects should be able to provide informed written consent (study participation informed consent form): Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Confirmed severe asthma diagnosis and treatment requirements according to American Thoracic Society(ATS)/European Respiratory Society (ERS) guidelines and Global Initiative for Asthma (GINA) 2023.
* Blood eosinophils ≥150cells/ul at screening visit or ≥300cells/ul the last 12 months.
* Patients with history ≥ 1 exacerbation the previous year under the treatment of high dose of inhaled corticosteroid(ICS)+LABA±LAMA or receiving oral/systemic corticosteroids at least 3 days. For subjects on maintenance oral corticosteroids, an exacerbation requiring oral corticosteroids was defined as the use of oral/systemic corticosteroids at least double the existing dose for at least 3 days.
* Meet requirements for biologic therapy with Benralizumab.

Exclusion Criteria:

* Asthma exacerbation, within 6 weeks prior to screening that required hospitalization or emergency room visit.
* Prior use of other biologics that has potential to interfere/ affect disease progression.
* Pregnant or nursing women, or women of child-bearing potential.
* History of malignancy of any organ system or any other serious co-morbidities defined by the treating physician.
* Patients with a history of conditions other than asthma that could result in elevated eosinophils (e.g. hypereosinophilic syndromes, Churg-Strauss Syndrome, eosinophilic esophagitis).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in sub-basement membrane thickness | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment.
Change in airway smooth muscle area | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment.
Change in airway smooth muscle layer thickness | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment.
Change in submucosal eosinophil number | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment.
Change in epithelial integrity | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment.
Change in collagen thickness | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. Any improvement in this parameter will be measured as change from baseline compared to measurement after 1 year of treatment, measured by electron microscopy.

SECONDARY OUTCOMES:
Change of cytokine and protein levels | through study completion, 52 weeks
  To identify any possible biomarkers of response of non-responders versus super-responders in different biological fluids as peripheral blood and bronchial washing. The identification of clinical characteristics of non-responders and super-responders.
  Change from baseline compared to measurements after 6 months and after 1 year of benralizumab treatment.
Change in exacerbation rate | through study completion, 52 weeks
  Measurement of the change in exacerbation rate in each severe eosinophilic asthmatic patient under benralizumab treatment for 52 weeks of treatment.
Change in blood eosinophil levels | through study completion, 52 weeks
  Measurement of the change in blood eosinophil levels in each severe eosinophilic asthmatic patient under benralizumab treatment for 52 weeks of treatment.
dentification of clinical characteristics of response, change in Forced Expiratory Volume (FEV1) | through study completion, 52 weeks
  The identification of clinical characteristics of non-responders and super-responders. FEV1 change from baseline, before treatment initiation, compared to measurements every 3 months until 1 year of treatment. FEV1 is the maximal amount of air you can forcefully exhale in one second measured by spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Kalliopi Domvri, Dr, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Pulmonary Clinic, Aristotle University of Thessaloniki, George Papanikolaou Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
A reference of the published article will be shared here.
Supporting Information: Study Protocol, CSR
Time Frame: Starting 9 months after publication and ending 36 months following article publication.
Access Criteria: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For individual participant data meta-analysis, data will be shared. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided).

REFERENCES:
- [Result] Kuo CW, Liao XM, Huang YC, Chang HY, Shieh CC. Bronchoscopy-guided bronchial epithelium sampling as a tool for selecting the optimal biologic treatment in a patient with severe asthma: a case report. Allergy Asthma Clin Immunol. 2019 Nov 27;15:76. doi: 10.1186/s13223-019-0378-6. eCollection 2019. PMID 31798645
- [Result] Bara I, Ozier A, Tunon de Lara JM, Marthan R, Berger P. Pathophysiology of bronchial smooth muscle remodelling in asthma. Eur Respir J. 2010 Nov;36(5):1174-84. doi: 10.1183/09031936.00019810. PMID 21037369
- [Result] Rasmussen F, Taylor DR, Flannery EM, Cowan JO, Greene JM, Herbison GP, Sears MR. Risk factors for airway remodeling in asthma manifested by a low postbronchodilator FEV1/vital capacity ratio: a longitudinal population study from childhood to adulthood. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1480-8. doi: 10.1164/rccm.2108009. PMID 12045120
- [Result] Yancey SW, Keene ON, Albers FC, Ortega H, Bates S, Bleecker ER, Pavord I. Biomarkers for severe eosinophilic asthma. J Allergy Clin Immunol. 2017 Dec;140(6):1509-1518. doi: 10.1016/j.jaci.2017.10.005. PMID 29221581
- [Result] Siddiqui S, Bachert C, Bjermer L, Buchheit KM, Castro M, Qin Y, Rupani H, Sagara H, Howarth P, Taille C. Eosinophils and tissue remodeling: Relevance to airway disease. J Allergy Clin Immunol. 2023 Oct;152(4):841-857. doi: 10.1016/j.jaci.2023.06.005. Epub 2023 Jun 19. PMID 37343842
- [Result] Berair R, Hartley R, Mistry V, Sheshadri A, Gupta S, Singapuri A, Gonem S, Marshall RP, Sousa AR, Shikotra A, Kay R, Wardlaw A, Bradding P, Siddiqui S, Castro M, Brightling CE. Associations in asthma between quantitative computed tomography and bronchial biopsy-derived airway remodelling. Eur Respir J. 2017 May 1;49(5):1601507. doi: 10.1183/13993003.01507-2016. Print 2017 May. PMID 28461289